CLINICAL TRIAL: NCT01543542
Title: A Phase II Multi-institutional Study Assessing Simultaneous In-Field Boost Helical Tomotherapy for 1-3 Brain Metastases
Acronym: TOMOSIBII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, George Rodrigues, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-10-204; 16776 (Other: Research Ethics Board)
Record Dates: First submitted 2012-02-16; First posted 2012-03-05 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Metastasis to Brain of Primary Cancer
Keywords: 1-3 brain metastases from any primary cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation Therapy Treatment (Other): Whole Brain XRT 30Gy/10 fractions with Simultaneous Infield Boost of Brain Lesions to 60Gy
  Interventions: Radiation: Whole Brain XRT 30Gy/10 fractions with

INTERVENTIONS:
Radiation: Whole Brain XRT 30Gy/10 fractions with — 30 Gy of whole brain external beam radiation delivered in 10 fractions. Simultaneous in-field boost of brain lesions to 60 Gy.

SUMMARY:
Helical tomotherapy is a novel radiation treatment machine that combines two existing technologies: spiral radiotherapy treatments combined with simultaneous computed tomotherapy imaging of the body. This new machine can potentially allow radiation treatments to be focused more precisely, and delivered more accurately than with existing radiation machines. In this study, helical tomotherapy will be used to provide radiation treatments (whole brain radiotherapy, daily over 10 treatments) that are commonly used to treat cancer metastatic to the brain. In addition, the individual spots of cancer (metastases) in the brain will be treated to a higher dose (approximately 2 times higher) than the dose to the whole brain. The purpose of this study is to determine the effectiveness of whole brain radiation with lesion boosting with the helical tomotherapy machine.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of primary cancer
* Contrast enhanced MRI demonstrating 1-3 metastases within 6 weeks of enrollment
* Age greater than or equal to 18
* Karnofsky performance status greater than or equal to 70
* Patient available for subsequent follow-up appointments and testing as well as health-related quality of life questionnaires
* Anticipated survival (independent of the brain metastases) greater than 3 months
* Patient informed consent obtained
* Metastatic suitable for synchronous boost
* Extracranial disease controlled or to be treated

Exclusion Criteria:

* Underlying medical condition precluding adequate follow-up
* Prior cranial radiotherapy
* Concurrent cytotoxic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2010-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Overall survival | At approximately end of year 4 (study completion)
Local disease control rate at 6 months | At approximately 2.5 years
CNS disease control rate at 6 months | At approximately 2.5 years

SECONDARY OUTCOMES:
Assessment of RTOG versus RECIST versus Volumetric MRI criteria | At approximately end of year 4 (study completion)
Health related quality of life | At approximately end of year 4 (study completion)
Karnofsky performance status | AT approximately end of year 4 (study completion)
Mini mental status exam cognition | At approximately end of year 4 (study completion)
Acute toxicity | At approximately end of year 4 (study completion)
Late toxicity | At approximately end of year 4 (study completion)
Changes in MRI endpoints | Measured at baseline, and 3 months and 6 months post-treatment
  Assessment in changes of diffusional weighted imaging and magnetic resonance spectroscopy. Changes at 3 months post-treatment and 6 months post-treatment will be compared to baseline (pre-treatment).

CONTACTS AND LOCATIONS:
Overall Officials: George Rodrigues, MD, MSc, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute; Glenn Bauman, MD, Principal Investigator — London Regional Cancer Program of the Lawson Health Research Institute
Locations (5):
- Canada (5):
  - Alberta Health Services, Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Centre Hospitalier De L'Universite de Montreal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

REFERENCES:
- [Derived] Rodrigues G, Yartsev S, Tay KY, Pond GR, Lagerwaard F, Bauman G. A phase II multi-institutional study assessing simultaneous in-field boost helical tomotherapy for 1-3 brain metastases. Radiat Oncol. 2012 Mar 21;7:42. doi: 10.1186/1748-717X-7-42. PMID 22436144